CLINICAL TRIAL: NCT06588998
Title: Xengenic Cortical Membranes Versus Connective Tissue Graft With Coronally Advanced Flap for the Treatment of Peri-implant Soft Tissue Dehiscences: A Randomized, Controlled Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amr Anwar Mohamed Ellithy Yousef (Other)
Responsible Party: Sponsor-Investigator, Amr Anwar Mohamed Ellithy Yousef, assistant lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: peri-implant_1
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Immediate Implant; Connective Tissue Graft

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Xengenic Cortical membranes (Experimental)
  Interventions: Device: Xengenic Cortical membranes
- connective tissue graft (Active Comparator)
  Interventions: Procedure: connective tissue graft

INTERVENTIONS:
Device: Xengenic Cortical membranes — soft tissue surgery around dental implant dehiscence
  Other Names: Osteobiol ,flexible xenograft cortical sheet from Technoss,USA
  Arms: Xengenic Cortical membranes
Procedure: connective tissue graft — soft tissue surgery around dental implant dehiscence
  Arms: connective tissue graft

SUMMARY:
Peri-implant soft tissue dehiscences represent a common complication in implant dentistry, often leading to esthetic and functional challenges. Current treatment options, including Xengenic cortical membranes and connective tissue graft with coronally advanced flap, aim to promote soft tissue regeneration and improve clinical outcomes. However, there is a need for comparative studies to determine the optimal treatment modality for peri-implant soft tissue dehiscences.

DETAILED DESCRIPTION:
Aim: Comparing the effectiveness and patient outcomes of Xengenic cortical membranes versus connective tissue graft with coronally advanced flap for the treatment of peri-implant soft tissue dehiscences.

ELIGIBILITY:
Inclusion Criteria:

* Adults (20-50) years old. •peri-implant soft tissue dehiscence . •Thin gingival phenotype. •Optimal compliance as evidenced by no missing treatment appointments and positive attitude towards oral hygiene.

Exclusion Criteria:

* •Medically compromised patients and systemic conditions precluding implant and periodontal surgery. •Smokers, diabetics, pregnant or lactating women. •History of chemotherapy, radiotherapy in head and/or neck region. •Bisphosphonate therapy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
peri implant soft tissue thickness | six months

SECONDARY OUTCOMES:
pink esthetic score | six months

CONTACTS AND LOCATIONS:
Locations (1):
- TantaU, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided